CLINICAL TRIAL: NCT03913806
Title: FLuoresence Image Guided Surgery With A VEGF-targeted Tracer in Soft-tissue Sarcomas in Humans (FLASH)- A Feasibility Dose Escalation Study
Brief Title: FLuoresence Image Guided Surgery With A VEGF-targeted Tracer in Soft-tissue Sarcomas in Humans Approach With Bevacizumab-IRDye 800CW
Acronym: FLASH
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, G.M. van Dam, Professor of Surgery, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL61739.042.17
Record Dates: First submitted 2018-05-14; First posted 2019-04-12 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Intervention Model Description: phase I/II safety and dose-finding study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Bevacizumab-IRDye800CW
  Interventions: Drug: Bevacizumab-IRDye800CW

INTERVENTIONS:
Drug: Bevacizumab-IRDye800CW — dose finding:10mg; 25mg; 50mg

SUMMARY:
There is a need for better visualization of resection margins during surgery for soft tissue sarcoma. Optical molecular imaging of soft tissue sarcoma associated biomarkers is a promising technique to accommodate this need. The biomarker Vascular Endothelial Growth Factor (VEGF-A) is overexpressed in soft tissue sarcoma versus normal tissue and has proven to be a valid target for molecular imaging. VEGF-A can be targeted by the monoclonal antibody bevacizumab. Monoclonal antibodies can be labeled by the near-infrared (NIR) fluorescent dye IRDye800CW (800CW). The investigators hypothesize that bevacizumab-800CW accumulates in VEGF expressing cancer, enabling soft tissue sarcoma visualization using a NIR intraoperative camera system. In this pilot intervention study the investigators will determine the optimal dosage of bevacizumab-800CW (10, 25 or 50mg) to detect soft tissue sarcoma intraoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patients with soft tissue sarcoma who are scheduled to undergo surgical intervention with curative intent
* World Health Organization (WHO) performance score 0-2.
* Signed written informed consent

Exclusion Criteria:

* Medical or psychiatric conditions that compromise the patient's ability to give informed consent.
* Other invasive malignancy
* Pregnant or lactating women. Documentation of a negative pregnancy test must be available for woman of childbearing potential. Woman of childbearing potential are pre- menopausal women with intact reproductive organs and women less than two years after menopause.
* History of infusion reactions to bevacizumab or other monoclonal antibody therapies.
* Inadequately controlled hypertension with or without current antihypertensive medications
* Within 6 months prior to inclusion: myocardial infarction, Transient Ischemic Attack, Cerebral Vascular Accident, pulmonary embolism, uncontrolled chronic hepatic failure, unstable angina pectoris.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-12-22 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Tracer detection | up to 6 months
  Determine if accumulation of the fluorescent tracer bevacizumab-800CW can be detected with an intraoperative near infrared camera system to identify soft tissue sarcoma tissue during surgery

SECONDARY OUTCOMES:
Part 1: Dose finding | up to 6 months
  Identify two doses of the NIR antibody tracer conjugate that provide the best visualization of tumour tissue during surgery
Part 1: Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to 6 months
  To obtain information safety aspects of the tracer, side effects, adverse events (AE), serious adverse events (SAE) and suspected unexpected serious adverse reactions (SUSAR)
Part 2: Optimal dose | up to 6 months
  Define which of the two doses of conjugate identified in part 1 is the optimal dose for further development in a phase II trial

CONTACTS AND LOCATIONS:
Overall Officials: Gooitzen van Dam, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Damron TA. CORR Insights(R): What Are the Complication Rates and Factors Associated With Total Femur Replacement After Tumor Resection? Findings From the Japanese Musculoskeletal Oncology Group. Clin Orthop Relat Res. 2024 Apr 1;482(4):713-715. doi: 10.1097/CORR.0000000000002915. Epub 2023 Nov 7. No abstract available. PMID 37938137